CLINICAL TRIAL: NCT00096356
Title: A Randomized Double-Blind Placebo-Controlled Study Of Oral Coenzyme Q10 To Relieve Self-Reported Cancer Treatment Related Fatigue In Breast Cancer Patients
Brief Title: Coenzyme Q10 in Relieving Treatment-Related Fatigue in Women With Breast Cancer
Acronym: CoQ10
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: REBACCCWFU-97202; U10CA081851 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; Fatigue
Keywords: fatigue; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — coenzyme Q10; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 - CoQ10 & Vitamin E (Active Comparator): CoQ10 100mg capsule combined with Vitamin E 100 IU taken orally three times per day.
  Interventions: Dietary Supplement: CoQ10 & Vitamin E; Dietary Supplement: Placebo & Vitamin E
- Arm 2 - Placebo & Vitamin E (Placebo Comparator): Placebo-Vitamin E 100 mg/day in 3 doses
  Interventions: Dietary Supplement: Placebo & Vitamin E

INTERVENTIONS:
Dietary Supplement: CoQ10 & Vitamin E
  Other Names: CoenzymeQ10
  Arms: Arm 1 - CoQ10 & Vitamin E
Dietary Supplement: Placebo & Vitamin E

SUMMARY:
RATIONALE: Coenzyme Q10 is a vitamin that may be effective in relieving fatigue and depression in women who are undergoing chemotherapy for breast cancer.

PURPOSE: This randomized clinical trial is studying how well coenzyme Q10 works in relieving treatment-related fatigue in women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of coenzyme Q_10 on cancer treatment-related fatigue in women with breast cancer.

Secondary

* Determine the effect of this drug on overall quality of life of these patients.
* Determine the effect of this drug on depression in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to planned radiotherapy (yes vs no) and type of chemotherapy (anthracycline vs non-anthracycline). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning on the first day of chemotherapy treatment, patients receive oral coenzyme Q_10 and oral vitamin E three times daily.
* Arm II: Beginning on the first day of chemotherapy treatment, patients receive oral vitamin E and an oral placebo three times daily.

Treatment in both arms continues for 24 weeks in the absence of unacceptable toxicity.

Quality of life, fatigue, and depression are assessed at baseline and at 8, 16, and 24 weeks.

PROJECTED ACCRUAL: A total of 101-236 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* Hg > 11g/dl; supportive measures (erythropoietin, transfusion, iron therapy) should be utilized to assist with maintaining Hgb levels
* Total cholesterol > 160mg/dL.
* Female with primary cancer diagnosis (breast)
* Planned adjuvant chemotherapy (neoadjuvant chemotherapy is excluded)
* KPS > 60
* Bilirubin < 1.5 x ULN
* SGOT < 2.5 x ULN
* SGPT < 2.5 x ULN

Exclusion Criteria:

* Recent involuntary weight loss (> 5% of body weight in the past 3 months)
* Statin therapy - current or planned during study. Below is a list of some commonly used statin drugs.(Note: This is a helpful guide, not a complete list.)

  * Atorvastatin (Lipitor)
  * Cerivastatin
  * Fluvastatin (Lescol)
  * Lovastatin (Mevacor, Altocor, Advicor)
  * Mevastatin
  * Pravastatin (Pravachol)
  * Rosuvastatin
  * Simvastatin (Zocor)
* Current or planned use of the following medications for fatigue

  * Corticosteroids (intermittent use as part of chemotherapy regimen is allowed)
  * Amphetamines or other stimulants including methylphenidate (Ritalin)or modafinil (Provigil)
* Patients diagnosed with uncontrolled hypertension
* Breast cancer patients who are male
* Pregnant women are excluded from participation in this study. A Serum pregnancy test is required within 1 week of registration if the patient is a woman of childbearing potential.
* Anticoagulant therapy - current or planned during study (except for maintenance of catheter patency)
* Patients with uncontrolled thyroid dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2004-08-27 (Actual); Primary Completion 2009-08-31 (Actual); Study Completion 2009-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Lesser, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (31):
- United States (31):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Helen F. Graham Cancer Center at Christiana Hospital, Newark, Delaware
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MBCCOP - JHS Hospital of Cook County, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Heartland Research Consortium, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Southeastern Medical Oncology Center - Goldsboro, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Caldwell Memorial Hospital, Lenoir, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - South Carolina Cancer Specialists, PA at Hilton Head Medical Center, Hilton Head Island, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia

REFERENCES:
- [Background] Vitolins MZ, Case LD, Rapp SR, Lively MO, Shaw EG, Naughton MJ, Giguere J, Lesser GJ. Self-reported adherence and biomarker levels of CoQ10 and alpha-tocopherol. Patient Prefer Adherence. 2018 Apr 24;12:637-646. doi: 10.2147/PPA.S158682. eCollection 2018. PMID 29731611
- [Result] Lesser GJ, Case D, Stark N, Williford S, Giguere J, Garino LA, Naughton MJ, Vitolins MZ, Lively MO, Shaw EG; Wake Forest University Community Clinical Oncology Program Research Base. A randomized, double-blind, placebo-controlled study of oral coenzyme Q10 to relieve self-reported treatment-related fatigue in newly diagnosed patients with breast cancer. J Support Oncol. 2013 Mar;11(1):31-42. doi: 10.1016/j.suponc.2012.03.003. PMID 22682875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in medical clinics
Pre-assignment Details: There was no run-in period. Everyone enrolled was randomized.
Groups:
- Arm 1 - CoQ10 + Vitamin E: CoQ10 + Vitamin E 100mg/day in 3 doses
- Arm 2 - Placebo + Vitamin E: Placebo + Vitamin E 100mg/day in 3 doses
Period: Overall Study
Arm/Group | Arm 1 - CoQ10 + Vitamin E | Arm 2 - Placebo + Vitamin E
Started | 122 | 114
Completed | 78 | 61
Not Completed | 44 | 53
Not completed — Adverse Event | 11 | 9
Not completed — Physician Decision | 5 | 3
Not completed — Withdrawal by Subject | 17 | 23
Not completed — Lack of Efficacy | 1 | 0
Not completed — multiple reasons | 10 | 18

BASELINE CHARACTERISTICS:
Population: All participants
Groups:
- Arm 1 - CoQ10 & Vitamin E: CoQ10 plus Vitamin E 100mg/day in 3 doses
- Arm 2 - Placebo & Vitamin E: Placebo plus Vitamin E 100mg/day in 3 doses
- Total: Total of all reporting groups
Arm/Group | Arm 1 - CoQ10 & Vitamin E | Arm 2 - Placebo & Vitamin E | Total
Number analyzed (Participants) | 122 | 114 | 236
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 108 | 104 | 212
  >=65 years | 14 | 10 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (9.4) | 50.9 (9.7) | 51.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 114 | 236
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 3 | 1 | 4
  African-American | 15 | 11 | 26
  Caucasian | 104 | 102 | 206
Region of Enrollment [Number; unit: participants]
  United States | 122 | 114 | 236

OUTCOME MEASURES:

1. Primary Outcome: Effects of Coenzyme Q10 on Fatigue (as Measured by POMS-F) 24 Weeks Following Randomization
Description: POMS-F is the Profile of Mood States - fatigue scale. It ranges from 0 to 28; higher values indicate greater fatigue.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 - CoQ10 & Vitamin E | Arm 2 - Placebo & Vitamin E
Number analyzed (Participants) | 122 | 114
units on a scale | 6.96 (0.71) | 8.33 (0.79)
Statistical Analysis 1: Comparison: Arm 1 - CoQ10 & Vitamin E vs Arm 2 - Placebo & Vitamin E; Constrained repeated measures analysis of variance - constrained such that baseline fatigue was the same in both groups and unadjusted for any baseline covariates; Test type: Superiority or Other; p = 0.1815, Mixed Models Analysis — The a priori significance level was 0.05 for the primary outcome; there is no adjustment for multiple comparisons; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-3.39 to 0.64], Standard Error of Mean 1.03 — This is the estimate of the difference in arms (Co-Q10 minus placebo). Lower is better for this outcome

2. Secondary Outcome: Effects of Coenzyme Q10 on Quality of Life (as Measured by FACT-B) 24 Weeks Following Randomization
Description: FACT-B stands for Functional Assessment of Cancer Therapy - Breast. It measures quality of life. It is the total of the FACT subscales (emotional, social, functional, and physical) and the Breast subscale. Scores range from 0 to 144; higher scores reflect better overall quality of life.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 - CoQ10 & Vitamin E | Arm 2 - Placebo & Vitamin E
Number analyzed (Participants) | 122 | 114
units on a scale | 111.8 (1.81) | 109.8 (1.96)
Statistical Analysis 1: Comparison: Arm 1 - CoQ10 & Vitamin E vs Arm 2 - Placebo & Vitamin E; Constrained repeated measures analysis of variance - constrained to have equal means at baseline, unadjusted for other covariates; Test type: Superiority or Other; p = .3903, Mixed Models Analysis — 0.05 significance level; no multiple comparison adjustment; Mean Difference (Final Values) = 1.99, 95% CI 2-sided [-2.56 to 6.53], Standard Error of Mean 2.31 — This is the difference in treatment groups at 24 weeks (Co-Q10 minus Placebo). Higher is better for this outcome

3. Secondary Outcome: Effects of Coenzyme Q10 on Depression (as Measured by CES-D Short-form) 24 Weeks Following Randomization
Description: CES-D is the Center for Epidemiologic Studies Depression Form. It consists of 20 questions. The total score ranges from 0 to 60. Higher scores indicate greater depression.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Arm 1- CoQ10 & Vitamin E: CoQ10 100mg capsule combined with Vitamin E 100 IU taken orally three times per day.
Arm/Group | Arm 1- CoQ10 & Vitamin E | Arm 2 - Placebo & Vitamin E
Number analyzed (Participants) | 122 | 114
units on a scale | 11.7 (0.96) | 12.4 (1.05)
Statistical Analysis 1: Comparison: Arm 1- CoQ10 & Vitamin E vs Arm 2 - Placebo & Vitamin E; Constrained repeated measures analysis of variance, constrained such that the baseline means are equal, unadjusted of other covariates; Test type: Superiority or Other; p = .6014, Mixed Models Analysis — 0.05 significance level, unadjusted for multiple comparisons; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-3.25 to 1.88], Standard Error of Mean 1.31 — This is the difference between treatment groups at 24 weeks (Co-Q10 minus Placebo). Lower is better for this outcome

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: One month past the end of treatment
Arm/Group | Arm 1 - CoQ10 & Vitamin E | Arm 2 - Placebo & Vitamin E
Serious Adverse Events (participants affected / at risk) | 22/100 | 15/93
Other Adverse Events (participants affected / at risk) | 89/100 | 84/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - CoQ10 & Vitamin E (N=100) | Arm 2 - Placebo & Vitamin E (N=93)
ANC (Blood and lymphatic system disorders) | 11 (12) | 4 (4)
WBC (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
allergic reaction (General disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 3 (4)
fever (General disorders) | 2 (2) | 1 (1)
hypotension (Cardiac disorders) | 1 (1) | 0 (0)
ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
infection (Infections and infestations) | 2 (2) | 3 (4)
pain (General disorders) | 1 (1) | 2 (3)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
L vent sy d (Cardiac disorders) | 0 (0) | 1 (1)
abd pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
chest pain (Cardiac disorders) | 0 (0) | 1 (1)
hot flashes (General disorders) | 0 (0) | 2 (4)
nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
headache (General disorders) | 1 (1) | 0 (0)
insomnia (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - CoQ10 & Vitamin E (N=100) | Arm 2 - Placebo & Vitamin E (N=93)
alopecia (General disorders) | 8 (16) | 11 (19)
anorexia (General disorders) | 11 (13) | 5 (7)
arthralgia (General disorders) | 6 (10) | 2 (3)
constipation (General disorders) | 13 (18) | 5 (7)
cough (General disorders) | 1 (1) | 6 (8)
diarrhea (General disorders) | 13 (17) | 17 (22)
dizziness (General disorders) | 13 (15) | 14 (15)
edema (General disorders) | 4 (4) | 10 (13)
fatigue (General disorders) | 48 (83) | 47 (80)
fever (General disorders) | 2 (2) | 5 (5)
headache (General disorders) | 16 (23) | 23 (31)
heartburn (General disorders) | 30 (48) | 27 (31)
hot flashes (General disorders) | 5 (6) | 7 (9)
infection (General disorders) | 4 (6) | 5 (5)
insomnia (General disorders) | 34 (53) | 26 (44)
irritability (General disorders) | 13 (16) | 13 (21)
mucositis (General disorders) | 11 (12) | 6 (7)
myalgia (General disorders) | 5 (5) | 5 (7)
nausea (General disorders) | 59 (75) | 52 (71)
neuropathy (General disorders) | 13 (19) | 10 (15)
pain (General disorders) | 15 (22) | 13 (20)
rash (General disorders) | 12 (15) | 19 (27)
tachycardia (General disorders) | 1 (1) | 5 (5)
vomiting (General disorders) | 9 (9) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No